CLINICAL TRIAL: NCT03093818
Title: PREemptive Pharmacogenomic Testing for Preventing Adverse Drug REactions
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J.J.Swen (Other)
Collaborators: University of Liverpool (Other); Medical University of Vienna (Other); Centro di Riferimento Oncologico - Aviano (Other); Andaluz Health Service (Other Government); University of Patras (Other); University of Ljubljana (Other); Karolinska Institutet (Other); The Golden Helix Foundation (Unknown); Royal Dutch Pharmacists Association (KNMP) (Unknown); Bio.Logis Genetic Information Management (Unknown); University Paul Sabatier of Toulouse (Other); Uppsala University (Other); Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); Federal Institute for Drugs and Medical Devices (Unknown); St. Antonius Hospital (Other)
Responsible Party: Sponsor-Investigator, J.J.Swen, Associate Professor of Pharmacogenetics, Section Chair Laboratory, Department of Clinical Pharmacy and Toxicology, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 668353 (U-PGx)
Record Dates: First submitted 2017-03-06; First posted 2017-03-28 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Adverse Drug Reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A 10% random sample will be re-assessed for causality and severity of recorded ADE will by a second independent, blinded (unaware of patient allocation) assessor.
  Drug-genotype association of the ADE as per the Dutch Pharmacogenomics Working Group guideline will be assessed by a blinded review committee
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacogenomic testing arm (Experimental): 4,050 patients will provide a DNA sample. A pharmacogenomic test is performed. Results of this test are incorporated in the (electronic) medical record and combined with a clinical decision support system. Physicians and pharmacists may choose to use these results to guide drug and dose selection as per the Dutch Pharmacogenomics Working Group guidelines. Patients will receive a "Safety-Code card" containing their personal pharmacogenomics results, which can be used by other physicians or pharmacists during subsequent prescriptions.
  Interventions: Other: Pharmacogenomic testing
- Standard of care arm (No Intervention): 4,050 patients will provide a DNA sample. However, no pharmacogenomic test is performed until the study is completed. Physicians and pharmacists will prescribe and dispense drugs routinely, without using pharmacogenomic test results to guide drug and dose selection. Patients will receive a mock "Safety-Code card", which does not contain personal pharmacogenomics results.

INTERVENTIONS:
Other: Pharmacogenomic testing — The pharmacogenomic panel to be used incorporates 48 genetic variants for the following 13 "pharamacogenes": CYP2B6 (cytochrome P450), CYP2C19, CYP2C9, CYP2D6,CYP3A4, DPYD (dihydropyrimidine dehydrogenase), FVL (factor five Leiden), HLA-B (human leukocyte antigen), NUDT15 (Nudix hydrolase), SLCO1B1 (solute carrier organic anion transporter), TPMT (thiopurine methyltransferase), UGT1A1 (UDP-glucuronosyltransferase), and VKORC1 (vitamin K epoxide reductase complex).
  Arms: Pharmacogenomic testing arm

SUMMARY:
PREPARE is an international, prospective, multi-center, open, randomized, cross-over implementation study assessing the impact of pre-emptive pharmacogenomic testing, of a panel of actionable pharmacogenomic variants, on adverse event incidence. Additional outcomes include, healthcare expenditure, process indicators for implementation and provider adoption of pharmacogenomics.

DETAILED DESCRIPTION:
Pre-emptive pharmacogenomic testing will be implemented in clinical sites across seven European countries (United Kingdom, The Netherlands, Austria, Greece, Slovenia, Italy and Spain). The 36-month study is split into two (19 and 18-month) time-blocks. The participating countries are randomized to start with either implementing pharmacogenomics guided prescribing or with standard of care in the first block. In the pharmacogenomics guided prescribing arm, results of the pharmacogenomic test will be incorporated in the (electronic) medical record and may be used by physicians and pharmacists to guide drug and dose selection for 39 routinely prescribed drugs, as per the Dutch Pharmacogenomics Working Group guidelines. In the standard of care arm, patients will not receive pharmacogenomic testing. After this 19-month block, the countries switch to implementing the opposite strategy and will recruit new patients for a period of 18 months.

Patients are eligible for participation when they receive a first prescription for one or more of 39 drugs for which a Dutch Pharmacogenomic Working Group guideline is available (acenocoumarol, amitriptyline, aripiprazole, atomoxetine, atorvastatin, azathioprine ,capecitabine, citalopram, clomipramine, clopidogrel, codeine, doxepin, efavirenz, escitalopram, flecainide, flucloxacillin, fluorouracil, haloperidol, imipramine, irinotecan, mercaptopurine, metoprolol, nortryptiline, paroxetine, phenprocoumon, phenytoin, pimozide, propafenon, sertraline, simvastatin, tacrolimus, tamoxifen, tegafur, thioguanine, tramadol, venlafaxine, voriconazole, warfarin or zuclopenthixol). All patients will be followed for a minimum of three months and a maximum of 18 months. In total, 8,100 patients will be recruited; 4,050 will receive pharmacogenomic testing, and 4,050 will receive standard of care. Each implementation site will concentrate on, but is not limited to, recruiting patients within a specific therapeutic area. Therapeutic areas include primary care, general medicine, cardiology, oncology, psychiatry, neurology, and transplantation. It is hypothesized that implementing pharmacogenomics guided drug and dose selection will decrease incidence of clinically relevant adverse drug reactions by 30% (from 4% to 2.8% among those with actionable drug-gene interactions).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years old
* Subject must receive a first prescription (meaning no known prescription for this drug in the preceding 12 months) for one or more of 42 drugs, for which a Dutch Pharmacogenomic Working Group guideline is available, which is prescribed to them in routine care
* Subject is able and willing to take part and be followed-up for at least 12 weeks
* Subject is able to donate blood or saliva
* Subject has signed informed consent
* The study limit of enrolment (200 per arm, per 18-month block) for that drug has not been reached

Exclusion Criteria:

* Subject has previous (direct-to-consumer, or clinical) genetic testing for a gene important to the drug of inclusion
* Subject is pregnant or lactating
* Subject has a life expectancy estimated to be less than three months by treating clinical team
* Duration of the drug of inclusion total treatment length is planned to be less than seven consecutive days. A drug whose route of administration changes during the first seven days (e.g. intravenous to oral flucloxacillin) but whose total treatment duration is seven days or longer, is still eligible.
* For inpatients: hospital admission is expected to be less than 72 hours
* Subject is unable to consent to the study
* Subject is unwilling to take part
* Subject has no fixed address
* Subject has no current general practitioner
* Subject is, in the opinion of the Investigator, not suitable to participate in the study
* Subject has existing impaired hepatic or renal function for which a lower dose or alternate drug selection are already part of current routine care. This would not apply to any drugs specifically given to manage liver/renal impairment/transplantation.
* Subject has an estimated glomerular filtration rate (MDRD) of less than 15 ml/min per 1,73m2 in a subject with a functioning graft
* Subject has advanced liver failure (stage Child-Pugh C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6950 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of a clinically relevant adverse drug reaction which is caused by the drug of inclusion. For oncology patients only hematological toxicities (grade 4-5) and non-hematological toxicities (grade 3-5) will be considered clinically relevant. | 12 weeks
  Defined as an adverse drug reaction which is causally related to the drug of inclusion (definite, probable or possible), clinically relevant (CTCAE Grade 2,3,4 or 5) and associated with a drug-genotype interaction (as per the Dutch Pharmacogenomics Working Group guidelines)

SECONDARY OUTCOMES:
Physician and pharmacist adherence to Dutch Pharmacogenomics Working Group guidelines | 18 months
  Defined as adhering to the guidelines or not adhering to the guidelines
Healthcare expenditure related to adverse events | 18 months
  Any costs made as a result of an adverse event
Incidence of drug discontinuation due to an adverse event | 18 months
  Related to the drug of inclusion
Incidence of discontinuation due to lack of efficacy | 18 months
  Related to the drug of inclusion
Quality of life | 18 months
  Time trade-off question
Incidence of dose adjustments | 18 months
  Related to the drug of inclusion
Attitudes towards and knowledge of pharmacogenomics | 18 months
  Composite outcome: a list of seven questions regarding pharmacogenomics

CONTACTS AND LOCATIONS:
Overall Officials: Jesse J. Swen, PharmD PhD, Principal Investigator — Leiden University Medical Center; Munir Pirmohamed, MB ChB(Hons) PhD, Principal Investigator — University of Liverpool; Gere Sunder-Plassmann, MD, Principal Investigator — Medical University of Vienna; Giuseppe Toffoli, MD, Principal Investigator — Centro di Riferimento Oncologico; Cristina Lucía Dávila Fajardo, PharmD PhD, Principal Investigator — Andaluz Health Service; George P. Patrinos, PhD, Principal Investigator — University of Patras; Vita Dolzan, MD PhD, Principal Investigator — University of Ljubljana
Locations (7):
- Medical University of Vienna, Vienna, Austria
- University of Patras, Pátrai, Greece
- Centro di Riferimento Oncologico, Aviano, Italy
- Leiden University Medical Center, Leiden, Netherlands
- University of Ljubljana, Ljubljana, Slovenia
- Servicio Andaluz de Salud, Granada, Spain
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data management plan has been written to comply to FAIR principles.
  Findable:
  We will indicate the existence of the data in our scientific publications and at our website (www.upgx.eu).
  Accessible:
  The datasets will not be made openly accessible, but will become available upon request after publications of the main paper by the U-PGx consortium.
  Interoperable:
  We will make use of standardized scores and standardized methodologies for example the star allele nomenclature and rs-numbering for genetic variants.
  Reusable:
  We do not intend to licence our data. A data dictionary is available for the entire eCRF.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The datasets will not be made openly accessible, but will become available upon request after publications of the main paper by the U-PGx consortium.
Access Criteria: Requests to re-use the data sets by third parties will be addressed to U-PGx Executive Board including the coordinator, i.e. Leiden University Medical Center, the Netherlands.
URL: https://cordis.europa.eu/project/id/668353/results

REFERENCES:
- [Derived] Habtemariam HD, Guchelaar HJ, Manson LEN, Swen JJ, Kant AC, Bohringer S. Reporting Adverse Drug Events: A Comparison of an Online Patient Tool Versus Telephone-Based Monitoring in Community Pharmacy Patients in the Netherlands. Drug Saf. 2025 Nov;48(11):1205-1214. doi: 10.1007/s40264-025-01571-4. Epub 2025 Jun 14. PMID 40517185
- [Derived] Roncato R, Bignucolo A, Peruzzi E, Montico M, De Mattia E, Foltran L, Guardascione M, D'Andrea M, Favaretto A, Puglisi F, Swen JJ, Guchelaar HJ, Toffoli G, Cecchin E. Clinical Benefits and Utility of Pretherapeutic DPYD and UGT1A1 Testing in Gastrointestinal Cancer: A Secondary Analysis of the PREPARE Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2449441. doi: 10.1001/jamanetworkopen.2024.49441. PMID 39641926
- [Derived] Swen JJ, van der Wouden CH, Manson LE, Abdullah-Koolmees H, Blagec K, Blagus T, Bohringer S, Cambon-Thomsen A, Cecchin E, Cheung KC, Deneer VH, Dupui M, Ingelman-Sundberg M, Jonsson S, Joefield-Roka C, Just KS, Karlsson MO, Konta L, Koopmann R, Kriek M, Lehr T, Mitropoulou C, Rial-Sebbag E, Rollinson V, Roncato R, Samwald M, Schaeffeler E, Skokou M, Schwab M, Steinberger D, Stingl JC, Tremmel R, Turner RM, van Rhenen MH, Davila Fajardo CL, Dolzan V, Patrinos GP, Pirmohamed M, Sunder-Plassmann G, Toffoli G, Guchelaar HJ; Ubiquitous Pharmacogenomics Consortium. A 12-gene pharmacogenetic panel to prevent adverse drug reactions: an open-label, multicentre, controlled, cluster-randomised crossover implementation study. Lancet. 2023 Feb 4;401(10374):347-356. doi: 10.1016/S0140-6736(22)01841-4. PMID 36739136
- [Derived] Psarias G, Iliopoulou E, Liopetas I, Tsironi A, Spanos D, Tsikrika A, Kalafatis K, Tarousi D, Varitis G, Koromina M, Siamoglou S, Patrinos GP. Development of Rapid Pharmacogenomic Testing Assay in a Mobile Molecular Biology Laboratory (2MoBiL). OMICS. 2020 Nov;24(11):660-666. doi: 10.1089/omi.2020.0168. Epub 2020 Oct 16. PMID 33064577
- See also: Ubiquitous Pharmacogenomics (U-PGx) Consortium Official Website — http://upgx.eu/

DOCUMENTS (2):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT03093818/Prot_002.pdf
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03093818/SAP_001.pdf